CLINICAL TRIAL: NCT02762929
Title: A Phase 2, Randomized, Controlled, Multicenter, Evaluation of the Efficacy and Safety of Locally Administered HTX-011, HTX-002, or HTX-009 for Postoperative Analgesia Following Bunionectomy
Brief Title: Evaluation of the Efficacy and Safety of Locally Administered HTX-011 for Postoperative Analgesia Following Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTX-011-C2016-208
Record Dates: First submitted 2016-05-02; First posted 2016-05-05 (Estimated); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Pain; Bunions
Keywords: Analgesia; Bunionectomy
MeSH Terms: conditions — Pain, Postoperative; Bunion; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (11):
- HTX-011A: 200 mg (Experimental): HTX-011A (bupivacaine/meloxicam), 200 mg/6 mg via injection.
  Interventions: Drug: HTX-011A
- HTX-011B: 30 mg (Experimental): HTX 011B (bupivacaine/meloxicam), 30 mg/0.9 mg via injection.
  Interventions: Drug: HTX-011B
- HTX-011B : 60 mg (Experimental): HTX-011B (bupivacaine/meloxicam) 60 mg/1.8 mg via injection or instillation.
  Interventions: Drug: HTX-011B
- HTX-011B: 120 mg (Experimental): HTX- 011B (bupivacaine/meloxicam), 120 mg/3.6 mg via injection or instillation.
  Interventions: Drug: HTX-011B
- HTX-011B: 200 mg (Experimental): HTX- 011B (bupivacaine/meloxicam), 200 mg/6 mg via injection.
  Interventions: Drug: HTX-011B
- Bupivacaine HCI (Active Comparator): Bupivacaine HCI, 50 mg via injection.
  Interventions: Drug: Bupivacaine HCl
- Saline Placebo (Active Comparator): Saline placebo via injection.
  Interventions: Biological: Saline Placebo
- HTX-002, 60 mg (Experimental): HTX- 002, 60 mg via injection.
  Interventions: Drug: HTX-002
- HTX-002, 120 mg (Experimental): HTX-002, 120 mg via injection.
  Interventions: Drug: HTX-002
- HTX-002, 200 mg (Experimental): HTX-002, 200 mg via injection.
  Interventions: Drug: HTX-002
- HTX-009 (Experimental): HTX-009, 3.6 mg via injection.
  Interventions: Drug: HTX-009

INTERVENTIONS:
Drug: HTX-011A — HTX-011A (bupivacaine/meloxicam), via injection.
  Arms: HTX-011A: 200 mg
Biological: Saline Placebo — Saline placebo via injection.
  Arms: Saline Placebo
Drug: HTX-011B — HTX-011B (bupivacaine/meloxicam), via injection or instillation.
  Arms: HTX-011B : 60 mg; HTX-011B: 120 mg; HTX-011B: 200 mg; HTX-011B: 30 mg
Drug: HTX-002 — HTX-002, via injection.
  Arms: HTX-002, 120 mg; HTX-002, 200 mg; HTX-002, 60 mg
Drug: Bupivacaine HCl — Bupivacaine HCI, via injection.
  Arms: Bupivacaine HCI
Drug: HTX-009 — HTX-009, via injection.
  Arms: HTX-009

SUMMARY:
A Phase 2, Randomized, Controlled, Multicenter, Evaluation of the Efficacy and Safety of Locally Administered HTX-011 for Postoperative Analgesia Following Bunionectomy

DETAILED DESCRIPTION:
This study includes multiple formulations for formulation selection of the fixed-combination product and for the factorial design assessment of the contribution of each component. HTX-011A is the second formulation studied (HTX-011-49). HTX-011B is the final formulation studied (HTX-011-56), which was also included in subsequent Phase 2b and Phase 3 studies. For the factorial design assessment, HTX-002, a bupivacaine-only formulation in the same HTX-011 proprietary polymer, and HTX-009, a meloxicam-only formulation in the same HTX-011 proprietary polymer, were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female 18 years of age or older
2. Female subjects are eligible only if all of the following apply:

   1. Not pregnant (female subject of child bearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy test before surgery)
   2. Not lactating
   3. Not planning to become pregnant while participating in the study
   4. Be surgically sterile; or be at least two years post-menopausal; or have a monogamous partner who is surgically sterile; or be practicing double-barrier contraception; or practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity); or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the FDA for greater than 2 months prior to screening visits and commits to the use of an acceptable form of birth control for the duration of the study and for 30 days from completion of the study
3. Male subjects must be surgically sterile (biologically or surgically) or commit to the use of a reliable method of birth control for the duration of the study until at least 1 week after the administration of study medication
4. Be scheduled to undergo a primary unilateral first metatarsal bunionectomy repair, without collateral procedures, under regional anesthesia
5. Subject has not had a contralateral bunionectomy in the non-study foot in the past 3 months
6. Have the ability and be willing to comply with the study procedures.
7. Must be able to understand study procedures and give informed consent for the conduct for all study procedures, using an IRB approved consent form

Exclusion Criteria:

1. Unwilling to sign informed consent or not willing or able to complete all study procedures
2. Have a contraindication or be allergic to any medication to be used during the trial period
3. Have clinically significant cardiac abnormalities that, in the opinion of the investigator, would pose a health risk to the subject
4. Have American Society of Anesthesiologists (ASA) Physical Status classification system category ≥4
5. Have clinically significant renal or hepatic abnormalities: for example, AST or ALT > 3x ULN, creatinine > 2x ULN
6. Have another pre-existing painful condition that may confound pain assessments
7. Have another surgery planned within 30 days of procedure
8. Have a known or suspected history of alcohol or drug abuse, or a positive drug screen
9. Currently taking analgesics for a chronically painful condition, or has taken long acting opioids within 3 days of surgery, or taken any opioids within 24 hours of scheduled surgery for this study
10. Subjects with documented sleep apnea or are on home continuous positive airway pressure (CPAP)
11. Subjects who are receiving oxygen therapy at the time of screening
12. Have participated in a clinical trial within 30 days of planned surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Anaheim, California
  - Bakersfield, California
  - Pasadena, Maryland
  - Houston, Texas
  - San Antonio, Texas

REFERENCES:
- [Derived] Ottoboni T, Quart B, Pawasauskas J, Dasta JF, Pollak RA, Viscusi ER. Mechanism of action of HTX-011: a novel, extended-release, dual-acting local anesthetic formulation for postoperative pain. Reg Anesth Pain Med. 2019 Dec 16:rapm-2019-100714. doi: 10.1136/rapm-2019-100714. Online ahead of print. PMID 31843865

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study HTX-011-208 included multiple study parts, various study drugs, formulations, and administration techniques. It was pre-specified in the SAP to pool different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. We pooled different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. However for Outcome Measures, different doses of study drugs were presented separately.
Groups:
- HTX-011A: HTX-011A (bupivacaine/meloxicam), 200 mg/6 mg via injection.
- HTX-011B: HTX-011B (bupivacaine/meloxicam), 30-200 mg/0.9-6 mg via injection or instillation.
- HTX-002: HTX-002, 60-200 mg via injection.
Period: Overall Study
Arm/Group | HTX-011A | HTX-011B | Bupivacaine HCI | Saline Placebo | HTX-002 | HTX-009
Started | 32 | 175 | 25 | 104 | 64 | 30
Completed | 31 | 172 | 25 | 101 | 64 | 30
Not Completed | 1 | 3 | 0 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — exclusionary medication disclosed late | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study HTX-011-208 included multiple study parts, various study drugs, formulations, and administration techniques. It was pre-specified in the SAP to pool different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. We pooled different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. However for Outcome Measures, different doses of study drugs were presented separately.
Groups:
- Total: Total of all reporting groups
Arm/Group | HTX-011A | HTX-011B | Bupivacaine HCI | Saline Placebo | HTX-002 | HTX-009 | Total
Number analyzed (Participants) | 33 | 174 | 25 | 104 | 64 | 30 | 430
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 149 | 23 | 86 | 56 | 26 | 368
  >=65 years | 5 | 25 | 2 | 18 | 8 | 4 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (13.86) | 50.4 (13.79) | 52.7 (11.81) | 50.0 (13.46) | 50.2 (12.51) | 49.9 (13.41) | 50.3 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 148 | 22 | 91 | 57 | 27 | 372
  Male | 6 | 26 | 3 | 13 | 7 | 3 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 50 | 5 | 28 | 26 | 10 | 128
  Not Hispanic or Latino | 24 | 124 | 20 | 76 | 38 | 20 | 302
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 174 | 25 | 104 | 64 | 30 | 430

OUTCOME MEASURES:

1. Primary Outcome: Mean Summed Pain Intensity (SPI) Score Over 24 Hours
Description: The SPI is derived by summing the pain intensity score weighted by the scheduled time duration. SPI0-24 will be calculated by summing the Pain intensity (PI) score at the relevant time points weighted by the scheduled time duration since the prior PI assessment as follows: SPI0-24= PI1+PI2+2*PI4+2*PI6+2*PI8+2*PI10+2*PI12+2*PI14+4*PI18+6*PI24. Min = 0 (if PI=0 at every time) and Max = 240 (if PI=10 at every time).
Time Frame: 0-24 hours
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- HTX-011B: 60 mg: HTX-011B (bupivacaine/meloxicam), 60 mg/1.8 mg via injection or instillation.
- HTX-011B: 120 mg: HTX-011B (bupivacaine/meloxicam), 120 mg/3.6 mg via injection or instillation.
- HTX-011B: 200 mg: HTX-011B (bupivacaine/meloxicam), 200 mg/6 mg via injection.
- Bupivacaine HCI: 50 mg: Bupivacaine HCI, 50 mg via injection.
- HTX-002, 60 mg: HTX-002, 60 mg via injection.
Arm/Group | HTX-011A: 200 mg | HTX-011B: 30 mg | HTX-011B: 60 mg | HTX-011B: 120 mg | HTX-011B: 200 mg | Bupivacaine HCI: 50 mg | Saline Placebo | HTX-002, 60 mg | HTX-002, 120 mg | HTX-002, 200 mg | HTX-009
Number analyzed (Participants) | 32 | 18 | 52 | 74 | 31 | 25 | 103 | 23 | 30 | 11 | 30
Units on a scale | 69.16 (43.092) | 96.83 (50.151) | 83.38 (46.226) | 85.70 (40.716) | 49.23 (40.781) | 118.16 (50.634) | 126.46 (47.785) | 112.00 (37.239) | 129.97 (45.897) | 107.82 (60.547) | 127.83 (49.196)

ADVERSE EVENTS:
Time Frame: 28 Days.
Description: Study HTX-011-208 included multiple study parts, various study drugs, formulations, and administration techniques. It was pre-specified in the SAP to pool different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. We pooled different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. However for Outcome Measures, different doses of study drugs were presented separately.
Groups:
- HTX-011A: HTX-011A (bupivacaine/meloxicam),200 mg/6 mg via injection.
- HTX-011B: HTX-011B (bupivacaine/meloxicam),30-200 mg/0.9-6 mg via injection or instillation.
Arm/Group | HTX-011A | HTX-011B | Bupivacaine HCI | Saline Placebo | HTX-002 | HTX-009
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/174 | 0/25 | 0/104 | 0/64 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/33 | 1/174 | 0/25 | 0/104 | 0/64 | 2/30
Other Adverse Events (participants affected / at risk) | 20/33 | 113/174 | 19/25 | 70/104 | 43/64 | 20/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HTX-011A (N=33) | HTX-011B (N=174) | Bupivacaine HCI (N=25) | Saline Placebo (N=104) | HTX-002 (N=64) | HTX-009 (N=30)
Impaired healing (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Post procedural cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HTX-011A (N=33) | HTX-011B (N=174) | Bupivacaine HCI (N=25) | Saline Placebo (N=104) | HTX-002 (N=64) | HTX-009 (N=30)
Cellulitis (Infections and infestations) | 3 | 5 | 0 | 1 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 4 | 0 | 1
Headache (Nervous system disorders) | 8 | 28 | 5 | 19 | 12 | 3
Dizziness (Nervous system disorders) | 5 | 10 | 2 | 8 | 4 | 3
Nausea (Gastrointestinal disorders) | 8 | 73 | 11 | 44 | 28 | 13
Vomiting (Gastrointestinal disorders) | 5 | 28 | 5 | 27 | 12 | 4
Constipation (Gastrointestinal disorders) | 2 | 17 | 1 | 20 | 8 | 4
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 4 | 2 | 1 | 4 | 3
Erythema (Skin and subcutaneous tissue disorders) | 3 | 18 | 2 | 3 | 9 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 9 | 0 | 1 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 8 | 4 | 7 | 6 | 0
Blister (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2 | 0 | 0
Feeling hot (General disorders) | 2 | 5 | 1 | 1 | 4 | 1
Oedema peripheral (General disorders) | 1 | 5 | 1 | 0 | 9 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 4 | 3 | 0 | 1 | 0 | 0
Eschar (Injury, poisoning and procedural complications) | 4 | 1 | 0 | 0 | 0 | 1
Hot Flush (Vascular disorders) | 2 | 1 | 0 | 2 | 1 | 0
Skin Warm (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT02762929/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT02762929/SAP_001.pdf